CLINICAL TRIAL: NCT06008223
Title: Renal Protective Effect and Clinical Analysis of Vitamin B6 in Patients With Sepsis
Brief Title: Clinical Analysis of Vitamin B6 in Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Huzhou (Other)
Responsible Party: Principal Investigator, Wen-Ming Feng, Principal investigator, The First People's Hospital of Huzhou
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHuzhou 001
Record Dates: First submitted 2023-06-14; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Sepsis; Vitamin B6; Kidney Injury; Inflammatory Response; Oxidative Stress Response
MeSH Terms: conditions — Sepsis | interventions — Vitamin B 6; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (vitamin B6) (Experimental)
  Interventions: Drug: vitamin B6
- control group (0.9% sodium chloride solution) (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: vitamin B6 — The Patients in experimental group were given vitamin B6 injection 300mg/d (100mg/2ml× 3) intravenous injection.
  Arms: experimental group (vitamin B6)
Drug: 0.9% sodium chloride solution — That in control group were injected with 0.9% sodium chloride solution 6 ml intravenously.
  Arms: control group (0.9% sodium chloride solution)

SUMMARY:
Methodology Patients A total of 128 patients with sepsis and AKI who were admitted to several centers including Huzhou first people's Hospital combined with Wuxing People's Hospital, Linghu people's Hospital and Nanxun people's Hospital from November 1, 2021 to October 31, 2022 were included in the study. And all patients were diagnosed by clinical examination, Diagnostic criteria sepsis was diagnosed according to the international Sepsis-3 for patients with suspected infection using the quickly Sepsis related organ failure assessment (qSOFA). The qSOFA score consists of only three criteria: Glasgow Coma Scale (GCS) <15, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥22/min. A qSOFA score of 2 or more points indicates suspected sepsis. Criteria for AKI was defined according to the Kidney Disease Improving Global Outcomes (KDIGO), by the presence of one of the following: ①Increase in SCr by ≥ 0.3mg/dl (≥26.5 μ mol/L) within 48h；② Renal impairment is known or increase in SCr by ≥50% within 7days; ③ Oliguria for ≥4 hours.

All patients were authorized by their families to sign informed consent, and the study was approved by the ethics committee of the hospital.

Inclusion criteria: ①18-65 years old; ② The hospital survival time was more than 48 hours, and the medical records were complete; ③There is no history of vitamin B6 use in the recent period of admission (within 2 weeks before admission).

Exclusion criteria: ①Patients with chronic renal insufficiency or renal failure in the past; ②Related renal injury caused by reasons other than sepsis; ③At the time of admission to ICU, there was cardiac failure or cardiogenic shock in combination with sepsis; ④Patients who use nephrotoxic drugs or contrast agents; ⑤Previous kidney transplantation; ⑥Patients with restrictive use of positive inotropic drugs (such as left ventricular outflow tract stenosis); ⑦Age<18 or>65; ⑧pregnant woman.

Treatment 128 patients were divided into experimental and control group by random number table method, 64 patients in each group. Both groups were given routine treatment of sepsis and corresponding treatment of primary disease. The Patients in experimental group were given vitamin B6 injection 300mg/d (100mg/2ml× 3) intravenous injection, the course of treatment is one week or until the patient dies. That in control group were injected with 0.9% sodium chloride solution 6 ml intravenously.

Assessment The general clinical data of the two groups were recorded, including age, sex, acute physiology and chronic health status scoring system II (APACHE II), qSOFA, and the constituent ratio of primary disease before treatment.

The inflammatory reaction indexes of the two groups were detected before and on the 7th day of treatment, including Interleukin 6 (IL-6), interleukin 8 (IL-8), tumor necrosis factor (TNF-α) and endothelin-1 (ET-1). After collecting 5ml of fasting elbow vein blood from two groups of patients, the serum was separated by centrifugation (centrifugation radius: 3cm, rotation speed: 2000r/min, time: 10min), and then detected by enzyme-linked immunosorbent assay (ELISA). ELISA kits for IL-6 (ab178013), IL-8 (ab214030), and TNF-a(ab181241) were purchased from abcam company. ELISA kit for ET-1 (K7429-100) was purchased from BioVision. All ELISA experiments were performed according to the kit instructions.

The oxidative stress response indexs of the two groups were detected before and on the 7th day of treatment, including superoxide dismutase (SOD), glutathione (GSH), malondialdehyde (MDA). The xanthine oxidase method is used to detect SOD, the DTNB method is used to detect GSH, and the thiobarbituric acid method is used to detect MDA.

The renal function indexs before and after treatment were detected before and on the 7th day of treatment, including the blood urea nitrogen (BUN) and serum creatinine (sCr) and renal resistance index (RRI). RRI was detected by ultrasound.

And the clinical data, including the rate of renal replacement therapy, ICU length of stay, total hospitalization expenses, and 28-d mortality, were recorded.

Statistical analysis All measurements were expressed as mean ± standard deviation (x ± s). And the counting datas were expressed in the form of percentage [n (%)]. The statistical SPSS 23.0 software were performed using the two samples t-test and adjusted chi-square test for the two groups. P-value,0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* The hospital survival time was more than 48 hours, and the medical records were complete;
* There is no history of vitamin B6 use in the recent period of admission (within 2 weeks before admission).

Exclusion Criteria:

* Patients with chronic renal insufficiency or renal failure in the past;
* Related renal injury caused by reasons other than sepsis;
* At the time of admission to ICU, there was cardiac failure or cardiogenic shock in combination with sepsis;
* Patients who use nephrotoxic drugs or contrast agents;
* Previous kidney transplantation;
* Patients with restrictive use of positive inotropic drugs (such as left ventricular outflow tract stenosis);
* Age<18 or>65;
* pregnant woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Inflammatory response index | before treatment
  The inflammatory reaction indexes of the two groups were detected . After collecting 5ml of fasting elbow vein blood from two groups of patients, the serum was separated by centrifugation (centrifugation radius: 3cm, rotation speed: 2000r/min, time: 10min), and then detected by enzyme-linked immunosorbent assay (ELISA).
Inflammatory response index | on the 7th day of treatment
  The inflammatory reaction indexes of the two groups were detected . After collecting 5ml of fasting elbow vein blood from two groups of patients, the serum was separated by centrifugation (centrifugation radius: 3cm, rotation speed: 2000r/min, time: 10min), and then detected by enzyme-linked immunosorbent assay (ELISA).
Oxidative stress response index | before treatment
  The oxidative stress response indexs of the two groups were detected. The xanthine oxidase method is used to detect SOD, the DTNB method is used to detect GSH, and the thiobarbituric acid method is used to detect MDA.
Oxidative stress response index | on the 7th day of treatment
  The oxidative stress response indexs of the two groups were detected. The xanthine oxidase method is used to detect SOD, the DTNB method is used to detect GSH, and the thiobarbituric acid method is used to detect MDA.
Renal function index | before of treatment
  The renal function indexs before treatment were detected before the 7th day of treatment.
Renal function index | on the 7th day of treatment
  The renal function indexs after treatment were detected on the 7th day of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-Ming Feng, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Lu WL, Feng WM, Xu W, Liu LH, He LM. RENAL PROTECTIVE EFFECT AND CLINICAL ANALYSIS OF VITAMIN B 6 IN PATIENTS WITH SEPSIS. Shock. 2024 Jun 1;61(6):841-847. doi: 10.1097/SHK.0000000000002329. Epub 2024 Apr 26. PMID 38691102